CLINICAL TRIAL: NCT03569553
Title: A Field Study for the Evaluation of AIGIV Clinical Benefit and Safety in the Treatment of Patients With Inhalational Anthrax in a Broad Exposure Event Scenario
Brief Title: A Field Study Evaluating Clinical Benefit and Safety of AIGIV (ANTHRASIL®) in Inhalational Anthrax Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Emergent BioSolutions (Industry)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: AX-003A
Record Dates: First submitted 2018-06-15; First posted 2018-06-26 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Inhalational Anthrax
Keywords: Anthrax; Bacillus anthracis; Inhalational anthrax; Bacterial infection; AIGIV; Anthrasil; Anthrax immune globulin; Anti toxin; Polyclonal antibodies
MeSH Terms: conditions — Inhalation anthrax; Anthrax; Bacterial Infections | interventions — Anthrax Immune Globulin Intravenous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AIGIV: Inhalational anthrax patients who have been administered AIGIV (ANTHRASIL®) as per licensed US prescribing information.
  Interventions: Drug: AIGIV

INTERVENTIONS:
Drug: AIGIV — Anthrax Immune Globulin Intravenous (Human)
  Other Names: ANTHRASIL®

SUMMARY:
This study will evaluate safety and clinical benefit of AIGIV used for treatment of patients with inhalational anthrax. This study will be implemented only in the event of a major anthrax exposure event. The study is designed to collect information on safety, clinical benefit (such as extent of anthrax illness and survival) and serum concentrations of AIGIV (for AIGIV pharmacokinetics) and anthrax toxins from inhalational anthrax patients treated with AIGIV.

DETAILED DESCRIPTION:
This study is a post-marketing requirement from the FDA to evaluate safety and clinical benefit of AIGIV administered to patients as part of their medical care after inhalational exposure to Bacillus anthracis. Study information (i.e. data on safety and clinical benefit evaluation of AIGIV up to Day 30 following administration) and patient samples (for assessment of AIGIV pharmacokinetics and anthrax toxin levels) will be collected (up to Day 7 following AIGIV administration) prospectively to the extent possible; however, due to logistical complexities that will likely occur during a mass anthrax exposure event, most data for this study will be collected retrospectively (including scavenged patient samples for assessment of serum AIGIV concentration and anthrax toxin levels). Therefore, both prospective and retrospective data collection are allowed in this study to maximize the amount of information obtained from inhalational anthrax patients who have been administered AIGIV.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed or suspected inhalational anthrax linked to an identified broad exposure scenario.
* Treatment with AIGIV.
* Informed consent/assent (as applicable).

Exclusion Criteria:

* There are no exclusion criteria for subjects enrolling in this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inhalational anthrax patients who have received AIGIV.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2027-05-30 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Assessment of AIGIV clinical benefit by overall mortality rate | Up to Day 30
  Mortality rate (incidence of death) in patients with confirmed diagnosis of inhalational anthrax treated with AIGIV

SECONDARY OUTCOMES:
Assessment of AIGIV clinical benefit by time from symptom onset to death | Up to Day 30
  Time from symptom onset to death in patients with confirmed diagnosis of inhalational anthrax treated with AIGIV
Assessment of AIGIV clinical benefit by mortality rate at Day 7 and Day 30 | Up to Day 30
  Difference in mortality rate at Day 7 and Day 30 after AIGIV administration to patients with confirmed diagnosis of inhalational anthrax
Assessment of AIGIV safety by incidence of serious adverse drug reactions and serious suspected adverse drug reactions | Up to Day 30
  Combined incidence of serious adverse drug reactions (ie, serious adverse events related to AIGIV administration) and serious suspected adverse drug reactions (ie, serious adverse events that occur during or within 24 hours following AIGIV administration) in individuals treated with AIGIV
Mortality rate stratified by number of AIGIV doses administered | Up to Day 30
  Number of deaths stratified by number of AIGIV doses (single versus multiple doses) in patients with confirmed diagnosis of systemic anthrax treated with AIGIV

OTHER OUTCOMES:
Cause-specific mortality rate | Up to Day 30
  Number of deaths assigned to a specific cause in patients with confirmed diagnosis of inhalational anthrax treated with AIGIV
Mortality rate stratified by AIGIV treatment time from symptom onset | Up to Day 30
  Number of deaths stratified by AIGIV treatment time from symptom onset (early versus late onset of symptoms) in patients with confirmed diagnosis of inhalational anthrax
Mortality rate stratified by acute physiologic assessment and chronic health evaluation (APACHE) II score at baseline | Up to Day 30
  Number of deaths stratified by APACHE II score at baseline in patients with confirmed diagnosis of inhalational anthrax treated with AIGIV
Duration of hospitalization | Up to Day 30
  Length of hospitalization in patients with confirmed diagnosis of inhalational anthrax treated with AIGIV
Duration of intensive care unit (ICU) hospitalization | Up to Day 30
  Length of ICU stay in patients with confirmed diagnosis of inhalational anthrax treated with AIGIV
Incidence of ICU hospitalization | Up to Day 30
  Number of patients with confirmed diagnosis of inhalational anthrax treated with AIGIV admitted to ICU
Duration of mechanical ventilation | Up to Day 30
  Length of mechanical ventilation in patients with confirmed diagnosis of inhalational anthrax treated with AIGIV
Evaluation of sequential organ failure assessment (SOFA) score | Up to Day 14
  Increase in SOFA score from baseline in patients with confirmed diagnosis of inhalational anthrax treated with AIGIV
Assessment of AIGIV pharmacokinetics | Up to Day 7
  Serum concentration of AIGIV over time in patients with confirmed diagnosis of inhalational anthrax treated with AIGIV to determine AIGIV pharmacokinetic parameters such as maximum serum concentration, area under the concentration versus time (i.e, level of AIGIV circulating over time) and clearance
Assessment of anthrax toxin levels (protective antigen and lethal factor) | Up to Day 7
  Levels of anthrax toxins (protective antigen and lethal factor) over time in patients with confirmed diagnosis of inhalational anthrax treated with AIGIV

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Essink, MD, Principal Investigator